CLINICAL TRIAL: NCT07207395
Title: A Study of Open-label Orally Administered JBI-802 Alone or in Combination With Pembrolizumab in Patients With Advanced NSCLC Tumors Harboring an STK11 Mutation
Brief Title: A Study of Orally Administered JBI-802 Alone or in Combination With Pembrolizumab for Patients With Non-small Cell Lung Cancer With an STK11 Mutation.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Christ Hospital (Other)
Responsible Party: Principal Investigator, Alexander Starodub, MD, PhD, The Christ Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-001
Record Dates: First submitted 2025-10-02; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Lung Cancer (NSCLC)
Keywords: STK11 Mutation; NSCLC; Lung Cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Monotherapy (Experimental): JBI-082 Single Agent
  Interventions: Drug: JBI-802
- Combination (Experimental): JBI-802 plus Pembrolizumab
  Interventions: Drug: JBI-802; Drug: Pembrolizumab

INTERVENTIONS:
Drug: JBI-802 — LSD1/HDAC6 Inhibitor
Drug: Pembrolizumab — PD-1
  Arms: Combination

SUMMARY:
The purpose of this study is to determine the overall safety and tolerability of JBI-802 as single agent and in combination with Pembrolizumab.

DETAILED DESCRIPTION:
This is a single site, open-label, study to define the safety profile and overall response rate (ORR) and duration of response (DOR) activity of JBI-802 alone and in combination with Pembrolizumab in participants with Non-Small Cell Lung Cancer harboring an STK11 mutation. Dose of study medication will be 10 mg orally once daily, 4 days on and 3 days off cycle. Dose of Pembrolizumab will be 200mg every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged ≥18 years at Screening.
2. Participants with a histologically confirmed diagnosis of locally advanced or metastatic NSCLC harboring an STK11 mutation.
3. Screening laboratory values:

   * Absolute neutrophil count (ANC) ≥1500 cells/mm3.
   * Platelet count ≥100,000 cells/mm3.
   * Total bilirubin ≤1.5×ULN. Patients with Gilbert's syndrome may be enrolled with up to 3.0xULN.
   * AST and ALT ≤2.5×ULN (unless liver metastases are present then up to 5×ULN is allowed).
   * Calculated creatinine clearance (CrCL) ≥40 mL/min calculated per Institutional standard.
   * Prothrombin time (PT) or activated partial thromboplastin time (aPTT)

     * 1.5×ULN if participant is not anticoagulated (Note: If participant is on anticoagulants, the participant must be on a stable dose for at least 2 weeks prior to study entry.
4. Must have at least one measurable lesion on CT scan or MRI per RECIST 1.1
5. Resolution of any clinically significant toxic effects of prior therapy to Grade 0 or 1 according to the NCI CTCAE, Version 5.0 (exception of alopecia and Grade 2 peripheral neuropathy, chronic Grade 2 endocrinopathies as a result of prior immunotherapy).
6. Eastern Cooperative Oncology Group (ECOG) performance status of ≤2.
7. Able to swallow oral medication.
8. Willing and able to give informed consent and comply with protocol requirements for the duration of the study.
9. Willingness to use contraception by a method that is deemed effective by the Investigator by both males and female participants of childbearing potential (post-menopausal women must have been amenorrheal for at least 12 months to be considered of non-childbearing potential) and their partners throughout the treatment period and for at least 3 months following the last dose of study drug.

Exclusion Criteria:

1. Treatment with systemic anticancer therapy or an investigational agent within 2 weeks or 5 half-lives, whichever is shorter, prior to start of study drug treatment.
2. Major surgery ≤21 days prior to starting study drug or has not recovered from adverse effects of such procedure.
3. Surgery (eg, stomach bypass) or medical condition that might significantly affect absorption of medicines (as judged by the Investigator).
4. Radiotherapy within 2 weeks prior to start of study drug treatment (palliative radiation or stereotactic radiosurgery within 7 days prior to start of study treatment). Participants must have recovered from all radiotherapy-related toxicities.
5. Known malignant central nervous system disease other than neurologically stable, treated brain metastases- defined as metastasis having no evidence of progression or hemorrhage for at least 4 weeks after treatment (including brain radiotherapy). Must be off any systemic corticosteroids for the treatment of symptomatic brain metastases for at least 14 days prior to enrollment.
6. Severe or unstable medical condition, such as congestive heart failure (New York Heart Association [NYHA] Class III or IV), ischemic heart disease, uncontrolled hypertension, uncontrolled diabetes mellitus, psychiatric condition, as well as an uncontrolled cardiac arrhythmia requiring medication (≥Grade 2, according to NCI CTCAE Version 5), myocardial infarction within 6 months prior to starting study treatment, or any other significant or unstable concurrent cardiac illness. Note: Stable chronic atrial fibrillation is allowed.
7. Congenital long QT syndrome or corrected QT interval by Fridericia (QTcF) interval >480 msec for males and females, respectively, at Screening.
8. History of other previous or concurrent cancer that would interfere with the determination of safety or efficacy assessment with respect to the qualifying solid tumor malignancy.
9. Live vaccines within 30 days prior to the first dose of JBI-802.
10. Glucocorticoids for any purpose other than to modulate symptoms from an event of clinical interest) or for use as a premedication in participants with a known history of an IV contrast allergy administered as part of CT radiography. Inhaled, intranasal, intraocular, topical, and intraarticular joint injections of steroids are permitted.
11. Use of strong inhibitors of cytochrome P450 3A (CYP3A) within 14 days or 5 half-lives (whichever is longer) or grapefruit juice or grapefruit containing products within 7 days prior to Cycle 1 Day 1.
12. Use of strong inducers of CYP3A within 14 days or 5 half-lives (whichever is longer) prior to Cycle 1 Day 1.
13. Use of strong inhibitors of cytochrome CYP2D6 within 14 days or 5 half-lives (whichever is longer) prior to Cycle 1 Day 1.
14. Use of strong inducers of CYP2D6 within 14 days or 5 half-lives (whichever is longer) prior to Cycle 1 Day 1.
15. Major active infection requiring parenteral antibiotics.
16. Known active human immunodeficiency viruses infection or active infection with hepatitis B or C.
17. Active gastrointestinal disease (eg, Crohn's disease, ulcerative colitis, or short gut syndrome) or other malabsorption syndromes that would reasonably impact drug absorption.
18. Acute illness within 14 days prior to IP dosing unless mild in severity and approved by the Principal Investigator.
19. Presence of active infection requiring antibiotics.
20. Pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the Screening Visit through 90 days after the last dose of trial treatment.
21. Current participation in another clinical study of an investigational agents. Simultaneous participation in observational studies is acceptable after Principal Investigator approval.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | Up to 28 days after last dose of study drug
  Characterized overall and by type, seriousness, relationship to study treatment, timing, and severity graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0
Investigator Assessed ORR | Up to 28 days from last dose of study drug
  Investigator-assessed overall response rate (ORR) indicated by stable disease, partial response or complete response and progression free survival (PFS) as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- The Christ Hospital, Cincinnati, Ohio, United States